CLINICAL TRIAL: NCT00799955
Title: Comparison of Efficacy and Side Effects of Intrathecal Morphine and TAP Block for Post-cesarean Analgesia
Brief Title: Comparing 2 Types of Pain Relief After Cesarean Delivery: Spinal Morphine and TAP Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H08-01726
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Cesarean Delivery
Keywords: Cesarean delivery; post-operative analgesia; TAP block; ultrasound

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Subjects will receive 100 micrograms of spinal morphine, at the time of spinal needle insertion (standard care at BCW). At the end of the case, one of two investigators, using ultrasound, will visualize the transversus abdominis plane. A capped needle will be pushed against the skin to mimic the pressure sensation of the TAP block. The needle will not break the skin and nothing will be injected in this control group. The procedure will then be repeated on the other side. A dressing will be applied on each side to blind the subject and researcher to which group she is in.
  Interventions: Procedure: Placebo block
- 2 (Active Comparator): No additional spinal medications will be given. At the end of the case, one of the two investigators, under sterile conditions, and using ultrasound, will visualize the tip of a blunt regional anaesthesia needle entering the transversus abdominis plane. After careful aspiration to exclude vascular puncture, 1.5mg/kg of 0. 5% ropivacaine (to maximum dose of 20 mls = 100mg on each side) will be injected, under vision, into the transversus abdominis plane, on each side. The subjects will still have spinal anesthesia of the abdomen and therefore will not feel needle insertion as sharp although most will have a sensation of pressure. A dressing will be applied over the needle's entry points.
  Interventions: Procedure: Ultrasound-guided TAP block

INTERVENTIONS:
Procedure: Placebo block — 100 micrograms of spinal morphine
  Arms: 1
Procedure: Ultrasound-guided TAP block — 1.5mg/kg of 0. 5% ropivacaine (to maximum dose of 20 mls = 100mg on each side) will be injected into the transversus abdominis plane, on each side
  Arms: 2

SUMMARY:
Summary Brief Summary Standard care for pain relief after cesarean delivery is spinal morphine. Spinal morphine may be unsuitable for patients having general anesthetic or prior morphine-related side effects and can be less effective in patients with morphine tolerance. An alternative is a TAP block where local anesthetic is deposited between the abdominal muscles consequently numbing the area and providing pain relief. The investigators believe a TAP block will provide equivalent pain relief to spinal morphine.

DETAILED DESCRIPTION:
Detailed Description In North America, the standard of care is neuraxial morphine. This is an effective analgesic, but can still cause problems with nausea, vomiting and itching. Spinal morphine may be unsuitable for patients who have had morphine-related side effects in the past and can be less effective in patients with morphine tolerance. It is also poorly suited for patients who have had a general anesthetic, as anesthesiologists do not routinely access the spinal space purely for analgesia. It is only when they are using the spinal route for surgical anesthesia, that they will also deposit morphine to provide pain relief after surgery.

The abdominal wall incision is an important contributor to pain following a cesarean delivery. The nerves supplying the anterior abdominal wall between the internal oblique and transversus abdominis muscles. By depositing local anesthetic solution between these muscles on each side, it is possible to block all these nerves and provide analgesia for the incision of the anterior abdominal wall. This is known as the transversus abdominis plane block or TAP block.

Studies have shown the TAP block to be useful for midline laparotomies for open prostatectomies, bowel resection and as rescue analgesia for abdominal surgery. There are two studies which look specifically at TAP block after cesarean delivery but none of them have compared it directly the current standard.

This study is a direct comparison of spinal morphine and TAP block. Obviously, adequate analgesia is of paramount importance to the patient and those caring for her. Studies to date indicate that the TAP block provides similar analgesia to spinal morphine in the early post-operative period. Therefore it would be a reasonable alternative for those patients who cannot have spinal morphine or who can not tolerate spinal morphine due to its side effects.

The primary objective will be to investigate whether the tranversus abdominis plane block provides equivalent analgesia post-cesarean delivery, as intrathecal morphine.

The secondary objective will be to determine whether there is a difference in post-operative abdominal scar pain, at three months post-surgery.

This study will be a prospective, randomized, placebo-controlled, double blinded study.

The study will involve two groups. Both groups will have spinal anesthesia for the surgery provided with 9-12 mg heavy bupivacaine and 10 mcg fentanyl.

1. Control group: standard care plus a placebo block.
2. Intervention group: no additional spinal medications will be given and an ultrasound-guided TAP Block will be given instead of the standard intrathecal morphine.

Standard post-cesarean analgesia and PONV orders will be resumed post-delivery.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean delivery under spinal anesthesia patients.
* >28 weeks gestation
* ASA 1 and 2 classification of health
* Mothers presenting to the assessment unit with ruptured membranes or in early stages of labour for whom a vaginal birth was not planned and who are therefore in need of urgent cesarean delivery.
* Able to read and understand English,
* Only patients expected to deliver before midday will be approached for participation in the trial to facilitate post-operative data collection.

Exclusion Criteria:

* Mothers in active labour
* ASA classification 3 or above
* Emergency cesarean delivery for fetal heart rate abnormalities
* Cesarean delivery under general anesthesia
* Maternal age <19
* BMI >40.
* Cesarean deliveries where a CSE is planned.
* Mothers with a history of drug allergy to morphine or to local anesthetics
* Mothers who are likely to deviate from standard postpartum analgesia protocol because of history of morphine tolerance or sensitivity.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Morphine equivalents used in the 24h post-delivery | 24 hours post operation

SECONDARY OUTCOMES:
Pain scores at rest, and with movement as assessed by verbal analogue score on arrival to recovery and at 2, 6, 10, and 24h post-spinal drug administration; post-operative nausea and vomiting scores, sedation score, presence or absence of itch; presence | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Roanne Preston, MD, FRCPC, Principal Investigator — University of British Columbia; Heather Loane, MBBS, B.Med.Sci, Study Director — University of British Columbia; Joanne Douglas, MD, FRCPC, Study Director — University of British Columbia; Simon Massey, MB BCh, MRCP, FRCA, Study Director — University of British Columbia; Jessica Tyler, BSc, Study Director — University of British Columbia
Locations (1):
- BC Women's Hospital Dept of Anesthesia, Vancouver, British Columbia, Canada